CLINICAL TRIAL: NCT01703065
Title: A Pilot Study of the Effects of Cabozantinib (XL184) on Bone Turnover and the Microenvironment in Men With Non-Metastatic and Metastatic Castration-Resistant Prostate Cancer
Brief Title: Cabozantinib in Men With Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed 2017 for low accrual. Last data for primary outcome on 02Feb2015.
Sponsor: University of Washington (Other)
Collaborators: Prostate Cancer Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Celestia Higano, Principal Investigator, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7819; NCI-2012-01898 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Adenocarcinoma of the Prostate; Castration-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
Keywords: Prostate cancer; Bone metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Two separate patient population arms (metastatic CRPC and non-metastatic CRPC) but both populations are given the same interventional treatment and the same safety assessments.
Masking Description: Treatment is open label and non-randomized. Split in to two patient populations - metastatic CRPC and non-metastatic CRPC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Cabozantinib in metastatic CRPC (Experimental): Metastatic CRPC patients to receive cabozantinib PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib
- Cabozantinib in non-metastatic CRPC (Experimental): Non-Metastatic CRPC patients to receive cabozantinib PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Given orally once a day
  Other Names: BMS-907351; Cometriq; XL184; cabozantinib-s-malate

SUMMARY:
This pilot clinical trial studies cabozantinib in treating men with castration-resistant prostate cancer. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
Primary Outcome Measure:

1. Change in urinary N-telopeptide (uNTX) from baseline to after 6 weeks of treatment with cabozantinib in men with non-metastatic CRPC.

   Secondary Outcome Measures:
2. Changes in serum markers of bone metabolism from baseline to after 6 weeks of treatment with cabozantinib. Markers of bone metabolism in blood include bone specific alkaline phosphatase, alkaline phosphatase, LDH.
3. Changes in biomarker expression in bone biopsy samples. To include MET, AKT, FASN and VEGFR2 expression and phosphorylation status (activation) in osteoblasts/osteoclasts and prostate cancer cells. Will also include changes in markers of apoptosis, proliferation, and angiogenesis.

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
INCLUSION CRITERIA

1. The subject has a proven histologic diagnosis of prostate adenocarcinoma, but may have undergone prior surgery and/or radiation.
2. The subject must currently have castration resistant prostate cancer defined as 2 serial rising PSAs with a castrate level of testosterone (<50 ng/dL).
3. A subject with non-metastatic CRPC may not have received prior chemotherapy unless in the neoadjuvant or adjuvant setting > 24 months ago and may not have received prior zoledronic acid or denosumab.
4. A subject with metastatic CRPC must have bone metastases accessible for biopsy by CT guidance.
5. The subject must be willing to undergo sequential biopsy of bone or bone metastases.
6. Subjects must have discontinued additional hormonal (eg bicalutamide, abiraterone, estrogen) therapy prior to the first dose of cabozantinib. No antiandrogen withdrawal period is required.
7. Subjects previously treated on another investigational agent must have a 2-week or more washout before starting cabozantinib, depending on the agent, toxicity profile, and half-life. However, such patients may begin tetracycline dosing after consent is signed.
8. Subjects who are currently on GnRH agonists or antagonist therapy must continue androgen suppression.
9. The subject is ≥18 years old on day of consent.
10. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1.
11. Organ and marrow function as follows:

    1. ANC ≥1500/mm3 without colony stimulating factor support.
    2. Platelets ≥100,000/mm3.
    3. Hemoglobin ≥9 g/dL.
    4. Total bilirubin ≤1.5 x the upper limit of normal (ULN). For subjects with known Gilbert's disease, bilirubin≤3.0 mg/dL.
    5. Serum albumin ≥2.8g/dL.
    6. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance >50 mL/min. The Cockcroft and Gault equation should be used: Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72).
    7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN.
    8. Lipase <2.0 × ULN and no radiologic or clinical evidence of pancreatitis.
    9. Serum testosterone level <50 ng/dL.
    10. Urine protein/creatinine (UPC) ratio ≤1.0 unless the patient has a neobladder.
    11. Serum phosphorus, magnesium, calcium and potassium ≥ lower limit of normal (LLN).
12. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
13. Sexually active subjects and their partners must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study.

EXCLUSION CRITERIA

1. The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (eg, cytokines or antibodies) within 3 weeks, or nitrosoureas/ mitomycin C within 6 weeks before the first dose of study treatment.
2. Prior treatment with cabozantinib and other met inhibitors.
3. Prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, or before the first dose of study treatment.
4. The subject has received radiation therapy:

   1. to the thoracic cavity or gastrointestinal tract within 3 months of the first dose of study treatment.
   2. to bone or brain metastasis within 14 days of the first dose of study treatment.
   3. to any other site(s) within 28 days of the first dose of study treatment.
5. The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment.
6. The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
7. The subject has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs.
8. The subject has a primary brain tumor.
9. The subject has active brain metastases or epidural disease (Note: Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment. Baseline brain scans are not required to confirm eligibility.)
10. The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test results at screening ≥ 1.3 x the laboratory ULN.
11. The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted.
12. The subject requires chronic concomitant treatment of strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's Wort). Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.asp; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
13. The subject has experienced any of the following:

    1. clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment.
    2. hemoptysis of ≥0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment.
    3. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment.
14. The subject has radiographic evidence of cavitating pulmonary lesion(s).
15. The subject has tumor in contact with, invading or encasing major blood vessels.
16. The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
17. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    a. Cardiovascular disorders including: i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening.

    ii. Concurrent uncontrolled hypertension defined as sustained BP > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days before the first dose of study treatment.

    iii. Any history of congenital long QT syndrome. iv. Any of the following within 6 months before the first dose of study treatment:
    * unstable angina pectoris
    * clinically-significant cardiac arrhythmias
    * stroke (including TIA, or other ischemic event)
    * myocardial infarction
    * thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study) b. Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including: i. Any of the following within 28 days before the first dose of study treatment:
    * intra-abdominal tumor/metastases invading GI mucosa
    * active peptic ulcer disease
    * inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
    * malabsorption syndrome ii. Any of the following within 6 months before the first dose of study treatment:
    * abdominal fistula
    * gastrointestinal perforation
    * bowel obstruction or gastric outlet obstruction
    * intra-abdominal abscess. Note: Complete resolution of an intraabdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months before the first dose of study treatment.

      c. Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy.

      d. Other clinically significant disorders such as: i. active infection requiring systemic treatment within 28 days before the first dose of study treatment ii. serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment iii. history of organ transplant iv. concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment v. history of major surgery as follows:
    * Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
    * Minor surgery within 1 months of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
18. The subject is unable to swallow tablets.
19. The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before Day 1 of Cycle 1. Note: if initial QTcF is found to be > 500 ms, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤500 ms, the subject meets eligibility in this regard.
20. The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.
21. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
22. For disease specific studies: The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment.
23. The subject has a known allergy to tetracycline.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2015-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celestia S Higano, MD, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Seattle Cancer Care Alliance/University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC
Started | 9 | 0
Completed | 8 | 0
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: 0 nmCRPC patients enrolled, so 0 nmCRPC patients analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 5
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 8 |  | 8
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 6 |  | 6
  More than one race | 0 |  | 0
  Unknown or Not Reported | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary N-telopeptide (uNTX) as a Marker of Bone Metabolism in Non-metastatic Patients
Description: Median percent change in Urinary N-Telopeptide from baseline compared to after 6 weeks of treatment with Cabozantinib in patients with non-metastatic prostate cancer.
Time Frame: Baseline and 6 weeks
Population: Of 9 total patients enrolled, 0 had non-metastatic CRPC, therefore this outcome was not analyzed.
Arm/Group | Cabozantinib in Non-metastatic CRPC
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Bone Specific Alkaline Phosphatase as a Marker of Bone Metabolism
Description: Median percent change in Bone Specific Alkaline Phosphatase from baseline compared to after 6 weeks of treatment with Cabozantinib.
Time Frame: Baseline and at 6 weeks
Population: Bone Specific Alkaline Phosphate was analyzed in blood samples from 8 patients with metastatic CRPC at baseline and following 6 weeks of treatment. 1 participant did not provide a 6 week sample, and was therefore excluded from this analysis. 0 participants were enrolled in the non-metastatic CRPC arm.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC
Number analyzed (Participants) | 8 | 0
percent change | 42.83 [-45.10 to 269.23] |

3. Secondary Outcome: Change in Alkaline Phosphatase as a Marker of Bone Metabolism
Description: Median percent change in Alkaline Phosphatase from baseline compared to after 6 weeks of treatment with Cabozantinib.
Time Frame: Baseline, 6 weeks
Population: Alkaline Phosphatase was analyzed in blood samples from 7 patients with metastatic CRPC at baseline and following 6 weeks of treatment. 2 participants did not provide a 6 week sample and were therefore excluded from this analysis. 0 participants were enrolled in the non-metastatic CRPC arm.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC
Number analyzed (Participants) | 7 | 0
percent change | 23.88 [-28.92 to 272.09] |

4. Secondary Outcome: Change in Lactic Acid Dehydrogenase (LDH) as a Marker of Bone Metabolism
Description: Median percent change in Lactic Acid Dehydrogenase (LDH) from baseline compared to after 6 weeks of treatment with Cabozantinib.
Time Frame: Baseline and at 6 weeks
Population: Lactic Acid Dehydrogenase (LDH) was analyzed in blood samples from 8 patients with metastatic CRPC at baseline and following 6 weeks of treatment. 1 participant did not provide a 6 week sample and was therefore excluded from this analysis. 0 participants were enrolled in the non-metastatic CRPC arm.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC
Number analyzed (Participants) | 8 | 0
percent change | 65.27 [12.59 to 120.07] |

5. Secondary Outcome: Changes in Biomarker Expression in Bone Biopsy Samples
Description: To include MET, AKT, FASN and VEGFR2 expression and phosphorylation status (activation) in osteoblasts/osteoclasts and prostate cancer cells. Will also include changes in markers of apoptosis, proliferation, and angiogenesis.
Time Frame: Baseline and at 6 weeks
Population: No nmCRCP patients enrolled, so no bone samples analyzed for this cohort. The purpose of biopsies in mCRPC cohort was to compare with those in nmCRPC cohort. Since no data to compare to, bone biopsy samples obtained were not analyzed. Only 1 patient with day 43 biopsy had specimen collected in both formalin and ethanol at baseline.
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each patient from first dose of study treatment through 30 days after the last dose of study treatment.
Description: Adverse events were recorded for patients in the metastatic arm. There were no patients enrolled in the non-metastatic arm.
Arm/Group | Cabozantinib in Metastatic CRPC | Cabozantinib in Non-metastatic CRPC
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/0
Other Adverse Events (participants affected / at risk) | 9/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib in Metastatic CRPC (N=9) | Cabozantinib in Non-metastatic CRPC (N=0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Refractory MultiFocal Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib in Metastatic CRPC (N=9) | Cabozantinib in Non-metastatic CRPC (N=0)
Fatigue (General disorders) | 9 | 0
Nausea (Gastrointestinal disorders) | 9 | 0
Dizziness (General disorders) | 3 | 0
Left hip pain (Injury, poisoning and procedural complications) | 2 | 0 — Pain from biopsy
Hypophosphatemia (General disorders) | 1 | 0
Dehydration (General disorders) | 4 | 0
Low back pain increased (Musculoskeletal and connective tissue disorders) | 2 | 0
Right shoulder pain - muscle (Musculoskeletal and connective tissue disorders) | 2 | 0
Dry mouth (General disorders) | 2 | 0
Dark colored urine (Renal and urinary disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Anorexia (Gastrointestinal disorders) | 8 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Hypokalemia (General disorders) | 3 | 0
Right hand neuropathy (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Weight loss (General disorders) | 4 | 0
Hypertension (Cardiac disorders) | 5 | 0
Mouth sore (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux (Gastrointestinal disorders) | 1 | 0
Chest pain, non-cardiac (General disorders) | 2 | 0
Laringeal inflammation (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Sacral pain (General disorders) | 1 | 0
ALT increased (Hepatobiliary disorders) | 4 | 0
AST increased (Hepatobiliary disorders) | 5 | 0
Dysgeusia (General disorders) | 4 | 0
Polyartralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flu-like symptoms (General disorders) | 1 | 0
Hemorrhoidal bleeding (General disorders) | 2 | 0
Right hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pelvis pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Seborrheic dermatitis, right ear (Skin and subcutaneous tissue disorders) | 1 | 0
Elevated TSH (Endocrine disorders) | 3 | 0
Rash, right groin (Skin and subcutaneous tissue disorders) | 1 | 0
Right scapular pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Weakness (General disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Headache (General disorders) | 2 | 0
Insomnia (General disorders) | 1 | 0
Night sweats (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Heart burn (Gastrointestinal disorders) | 1 | 0
Hoarseness (General disorders) | 3 | 0
Loose stools (Gastrointestinal disorders) | 2 | 0
GERD (Gastrointestinal disorders) | 4 | 0
Cervical and lumbar spine pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — post-traumatic
Left heel pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Telangiectasia cheeks (Vascular disorders) | 1 | 0
Hyperpigmented papules (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hand-Foot syndrome (General disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0
Runny nose (General disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Body aches (General disorders) | 1 | 0
increased triglycerides (Blood and lymphatic system disorders) | 1 | 0
Right upper arm bruising (General disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Bilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 1 | 0
Dry heaving (Gastrointestinal disorders) | 1 | 0
Hypercalcemia (General disorders) | 1 | 0
Pharingitis (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment goal was 34 evaluable patients. A total of 9 patients were consented and enrolled, 0 non-metastatic and 9 metastatic. Given that fewer patients enrolled than expected, some endpoints are not-evaluable or inconclusive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No